CLINICAL TRIAL: NCT00981929
Title: Development of Cocktail for Measuring the Activity of Important Cytochrome P450 Enzymes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unexpected non-serious adverse events
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Kim Brosen / Professor, University of Southern Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: AKF-375
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Cytochrome P450 Phenotype and Genotype Metrics
Keywords: CYP2D6; CYP2C9; CYP2C19; CYP1A2
MeSH Terms: interventions — Tramadol; Omeprazole; Losartan; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tramadol (Active Comparator): CYP2D6 metric
  Interventions: Drug: Tramadol
- Omeprazole, losartan, caffeine (Active Comparator): CYP2C19, CYP2C9 and CYP1A2 metrics
  Interventions: Drug: Omeprazole, losartan, caffeine
- Tramadol, omeprazole, losartan and caffeine (Active Comparator): CYP2D6, CYP2C19, CYP2C9 and CYP1A2 metrics
  Interventions: Drug: Tramadol, omeprazole, losartan, caffeine

INTERVENTIONS:
Drug: Tramadol — 50 mg single oral dose
  Arms: Tramadol
Drug: Omeprazole, losartan, caffeine — 20 mg omeprazole 25 mg losartan 200 mg caffeine
  Arms: Omeprazole, losartan, caffeine
Drug: Tramadol, omeprazole, losartan, caffeine — 50 mg tramadol 20 mg omeprazole 25 mg losartan 200 mg caffeine
  Arms: Tramadol, omeprazole, losartan and caffeine

SUMMARY:
The Cytochrome P450 enzymes are responsible for the metabolism of a wide range of drugs and other xenobiotics. Genetic variants of the encoding P450 genes have shown to influence the rate of metabolism of many clinically used drugs.

The drugs tramadol, omeprazole, losartan, quinidine and caffeine reflect the activity of CYP2D6 (tramadol), CYP2C19 (omeprazole), CYP2C9 (losartan), CYP1A2 (caffeine) and CYP3A4/5 (quinidine).

The aim of the study is to investigate if the cocktail of tramadol, omeprazole, losartan and caffeine can be used to simultaneously determine the activity of CYP2D6, CYP2C19, CYP2C9 and CYP1A2. Furthermore, will the natural occurring 4-beta-hydroxy-cholesterol in the blood be measured as a metric for CYP3A4/5.

The study is divided in two. First part will include 12 healthy volunteers and consists of three arms separated by at least one week. In the first arm 50 mg of tramadol will be ingested and urine will be collected for 8 hours. In the second arm 20 mg omeprazole, 25 mg losartan and 200 mg caffeine will be ingested followed by 8 hours urine collection and a blood sample 4 hours after administration of the drugs. In the last arm 50 mg of tramadol, 20 mg omeprazole, 25 mg losartan and 200 mg caffeine will be ingested followed by 8 hours urine collection and a blood sample 4 hours after administration of the drugs.

Metabolic ratios will be calculated based on urine and plasma concentrations of the drugs and the relevant metabolites. Relevant genetic variants of the cytochrome P450 encoding genes will be determined.

If the metabolic ratios of the drugs are not significantly different between the arms, Second part of the study will be conducted.

This part is identical with the last arm and will include a maximum of 400 healthy volunteers: 50 mg of tramadol, 20 mg omeprazole, 25 mg losartan and 200 mg caffeine will be ingested followed by 8 hours urine collection and a blood sample 4 hours after administration of the drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers,
* Written consent, AND
* Age 18-65 years old.

Exclusion Criteria:

* Daily medication,
* Alcohol abuse,
* Pregnancy, OR
* Breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-12 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic ratios | January 2011

SECONDARY OUTCOMES:
Genetic variants | January 2011

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Denmark, Clinical Pharmacology, Odense, Fyn, Denmark

REFERENCES:
- [Derived] Pedersen RS, Damkier P, Christensen MM, Brosen K. A cytochrome P450 phenotyping cocktail causing unexpected adverse reactions in female volunteers. Eur J Clin Pharmacol. 2013 Dec;69(12):1997-9. doi: 10.1007/s00228-013-1561-1. Epub 2013 Aug 6. PMID 23917460